CLINICAL TRIAL: NCT06962839
Title: A Randomised, Double-masked, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Oral BI 1815368 in Participants With Centre-involved Diabetic Macular Edema for 48 Weeks of Treatment (THULITE)
Brief Title: A Study to Test Whether BI 1815368 Helps People With an Eye Condition Called Diabetic Macular Edema
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1485-0018; U1111-1317-2206 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP)); 2024-520384-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Intervention Model Description: Participants in Cohort 1 will be randomised in a 1:1 ratio to placebo or BI 1815368 group.
  Once Cohort 1 is fully recruited, Cohort 2 will be randomised in a 1:1:1:1 ratio to placebo or BI 1815368 low/medium/high dose groups.
  There is no planned pause in recruitment between Cohort 1 and Cohort 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Treatment arm (Experimental)
  Interventions: Drug: BI 1815368
- Cohort 1: Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2: Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2: Treatment arm, low dose (Experimental)
  Interventions: Drug: BI 1815368
- Cohort 2: Treatment arm, medium dose (Experimental)
  Interventions: Drug: BI 1815368
- Cohort 2: Treatment arm, high dose (Experimental)
  Interventions: Drug: BI 1815368

INTERVENTIONS:
Drug: BI 1815368 — BI 1815368
  Arms: Cohort 1: Treatment arm; Cohort 2: Treatment arm, high dose; Cohort 2: Treatment arm, low dose; Cohort 2: Treatment arm, medium dose
Drug: Placebo — Placebo matching BI 1815368
  Arms: Cohort 1: Placebo arm; Cohort 2: Placebo arm

SUMMARY:
This study is open to adults 18 and older with an eye condition called diabetic macular edema. People are required to have a specific type of diabetic macular edema called centre-involved diabetic macular edema (CI-DME) to take part. The purpose of this study is to find out whether a medicine called BI 1815368 improves sight in people with CI-DME and to find the most suitable dose.

This study has 2 parts. In the first part, participants are put into 2 groups of equal size randomly, which means by chance. One group takes BI 1815368 tablets and the other group takes placebo tablets. Placebo tablets look like BI 1815368 tablets but do not contain any medicine. In the second part, participants are put into 4 groups of equal size randomly. 3 groups take different daily doses of the study medicine, BI 1815368, while 1 group takes placebo. All participants take tablets twice a day for about 11 months.

Participants are in the study for about 1 year. During this time, they visit the study site 16 times. At visits, doctors check the participant's vision and collect information on any health problems. They take detailed pictures of the eye. The changes over time are compared between the groups to see if the treatment works.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years of age
* Diagnosis of diabetes mellitus (DM) (type 1 or type 2), Haemoglobin A1C (HbA1c) <12% treated with stable medication for at least 30 days prior to Day 1; no already-set plans for major changes in DM medication (e.g. start of new medication) at the time of screening and baseline
* Centre-involved diabetic macular edema (CI-DME) confirmed on spectral domain optical coherence tomography (SD-OCT) with central subfield foveal thickness (CST) ≥320 µm for male and ≥305 µm for female participants in the study eye at screening
* Best corrected visual acuity (BCVA) visual acuity Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye between 24 and 78 (Snellen equivalent range 20/320 to 20/32) at screening Further inclusion criteria apply.

Exclusion criteria:

* Macular edema considered to be due to other causes than CI-DME in the study eye
* Proliferative diabetic retinopathy or iris neovascularisation (including the anterior chamber angle) in the study eye
* Any intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) treatment within 4 months before Day 1 (other than Vabysmo® or Eylea® HD), and within 6 months before Day 1 for Vabysmo® or Eylea® HD, and/or more than 4 prior IVT injections with anti-VEGF treatment in total in the study eye
* Any history of panretinal photocoagulation treatment, macular laser photocoagulation, vitreoretinal surgery, IVT or periocular corticosteroid treatment (within 12 months before Day 1), history of Iluvien® or Ozurdex® implants before Day 1, or topical steroid or NSAID treatment (within 30 days before Day 1)
* Active ocular inflammation of any history of intraocular inflammation within 1 year
* Aphakia or total absence of the posterior capsule; Yttrium aluminium garnet (YAG) laser capsulotomy in the study eye is permitted if more than 2 months prior to Day 1 Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Occurrence (yes/no) of a gain of ≥10 Early Treatment Diabetic Retinopathy Study (ETDRS) letters compared with baseline in the study eye at Week 48 | at baseline, at week 48
  With ETDRS letters, the number of letters a patient can correctly read on an ETDRS chart from a distance of 4 meters is measured.

SECONDARY OUTCOMES:
Occurrence (yes/no) of gain of ≥15 ETDRS letters compared with baseline in the study eye at Week 48 | at baseline, at week 48
  With ETDRS letters, the number of letters a patient can correctly read on an ETDRS chart from a distance of 4 meters is measured.
Occurrence (yes/no) of drug-related adverse events (AEs) over the treatment period through end of study (EoS) | up to 52 weeks
Absolute change from baseline of central subfield foveal thickness (CST) as measured by spectral domain optical coherence tomography (SD-OCT) in the study eye at Week 48 | at baseline, at week 48

CONTACTS AND LOCATIONS:
Locations (80):
- United States (23):
  - Win Retina, Arcadia, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Retinal Consultants Medical Group, Inc, Modesto, California
  - Doheny Eye Center UCLA Arcadia, Pasadena, California
  - Retina Consultants of San Diego, Poway, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - Colorado Retina Associates, Lakewood, Colorado
  - Advanced Research Institute, Pompano Beach, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Associated Vitreoretinal and Uveitis Consultants, Carmel, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Verum Research, LLC, Eugene, Oregon
  - Tennessee Retina, Nashville, Tennessee
  - Austin Research Center for Retina, PLLC, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Center Of Texas, Southlake, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
- China (5):
  - West China Hospital, Sichuan University, Chengdu
  - Shanghai General Hospital, Shanghai
  - The Fourth People's Hospital of Shenyang, Shenyang
  - Shijiazhuang People's Hospital, Shijiazhuang
  - Shanxi Eye Hospital, Taiyuan
- Czechia (7):
  - University Hospital Hradec Kralove (FNHK), Hradec Králové
  - University Hospital Ostrava, Ostrava-Poruba
  - Oftex s.r.o., Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Axon Clinical s.r.o., Prague
- Germany (5):
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Augenzentrum am St. Franziskus-Hospital Münster, Münster
- Hungary (8):
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associations Kft., Budapest
  - Budapesti Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - University of Debrecen, Debrecen
  - Nozologen Kft., Pécs
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Japan (9):
  - Asahikawa Medical University Hospital, Asahikawa-shi
  - Tokyo Medical University Hachioji Medical Center, Hachioji-shi
  - Kagawa University Hospital, Kita-gun
  - Kurume University Hospital, Kurume-shi
  - Shinshu University Hospital, Matsumoto-shi
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Nagoya City University Hospital, Nagayoga
  - Tokyo Women's Medical University Hospital, Tokyo
  - Juntendo University Urayasu Hospital, Urayasu-shi
- Poland (10):
  - Szpital Swietego Lukasza S. A., Bielsko-Biala
  - Oculomedica Sp. z o.o., Bydgoszcz
  - Clinical Medical Research Sp. z o.o., Katowice
  - Szpital Sw. Rozy Sp. z o.o., Krakow
  - Centrum Medyczne Dietla 19 Sp. z o.o., Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka-Lens Sp. z o.o., Olsztyn
  - Poznanskie Centrum Wzroku sp z o o, Poznan
  - Caminomed Sp. z o.o., Tarnowskie Góry
  - Eb Group Sp. z o.o., Warsaw
  - Warszawski Szpital Okulistyczny Sp. z o.o., Warsaw
- Slovakia (4):
  - F D Roosevelt University General Hospital Of Banska Bystrica, Banská Bystrica
  - Nemocnica s poliklinikou Trebisov a.s., Trebišov
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- United Kingdom (9):
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - Gloucestershire Royal Hospital, Gloucester
  - Northwick Park Hospital, Harrow
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - King's College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Sunderland Eye Infirmary, Sunderland
  - Southend University Hospital, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com